CLINICAL TRIAL: NCT02008630
Title: Animal-assisted Interventions in Health Promotion for Elderly With Dementia; Impact on Factors Related to Risk of Falls
Brief Title: Animal-assisted Interventions in Health Promotion for Elderly With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Life Sciences (Other)
Responsible Party: Principal Investigator, Camilla Ihlebæk, Professor, Norwegian University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012/1144-1
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Animal Assisted Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Animal-assisted activity (Experimental): 30 minutes group session with animal-assisted activity twice a week for 12 weeks in groups of 4-6 participants.
  Interventions: Other: Animal-assisted activity
- Animal-assisted therapy (Experimental): 30 minutes group session with animal-assisted therapy twice a week for 12 weeks in groups of 4-6 participants
  Interventions: Other: Animal-assisted therapy
- Control (No Intervention): Control group with treatment as usual

INTERVENTIONS:
Other: Animal-assisted activity
  Arms: Animal-assisted activity
Other: Animal-assisted therapy
  Arms: Animal-assisted therapy

SUMMARY:
The overall research aim of this study is to investigate changes in measures related to the risk of falls among elderly with dementia participating in animal-assisted interventions. Also relatives' experience of own and the elderly's situation during and after the intervention will be examined. The design will be a prospective and cluster randomized multicenter trial, but mixed-methods will be used to target different outcomes. The study population will be elderly (age above 65) at day care centers diagnosed with dementia, or having a cognitive deficit. The intervention will consist of 30 minutes sessions with animal-assisted activity or animal-assisted therapy two times a week for 12 weeks in groups of 4-6 participants. Control groups will receive treatment as usual. Research questions:

1. Is there an effect in use of ordinary and optional medication among elderly persons with dementia at day care centers participating in animal-assisted interventions compared to a control group?
2. Is there an effect on social interaction, quality of life, activeness and wellbeing among elderly persons with dementia at day care centers participating in animal-assisted interventions compared to a control group?
3. Is there an effect on balance among elderly persons with dementia at day care centers participating in animal-assisted therapy compared to animal-assisted activity or a control group?
4. Do relatives of elderly persons with dementia at day care centers experience a change in their own and the elderly's situation after the intervention compared with before the intervention started?

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of dementia or having a cognitive deficit measured as a score less than 25 on Mini-Mental State Examination.

Exclusion Criteria:

* Fear of dogs, dog allergy or need of wheel chair

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in Norwegian version of Berg balance test | Second last or last week before the intervention starts, after 4 and 8 weeks of the intervention, and first or second week after end of intervention. A follow-up measure 3 months after end of the intervention

SECONDARY OUTCOMES:
Change in Norwegian version of Quality of Life in Late-Stage Dementia (QUALID) | Second last or last week before the intervention starts, after 6 weeks of the intervention, and first or second week after end of intervention. A follow-up measure 3 months after end of the intervention

OTHER OUTCOMES:
Change in physical activity measured by Actigraphy | Second last or last week before the intervention starts, after 6 weeks of the intervention, and first or second week after end of intervention
  A device worn by the participants for one week at each time point of measure, night and day, measuring physical movement. Will be used to calculate physical activity during day time and sleep efficacy during the night.
Video recordings of two group session at each location | After two and ten weeks of the intervention
  The video recordings will be analyzed with respect to social interaction and group dynamics
Change in optional and ordinary medication | Second last or last week before the intervention starts, first or second week after the end of intervention. A follow-up measure 3 months after end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Ihlebæk, PhD, Principal Investigator — Norwegian University of Life Sciences
Locations (21):
- Norway (21):
  - Solgården Dagsenter, Asker
  - Lommedalen dagsenter, Bærum
  - Vallerhjemmet dagsenter, Bærum
  - Pålsetunet dagsenter, Fet
  - Fjerdingby dagsenter, Fjerdingby
  - Glemmen dagsenter, Fredrikstad
  - Tjølling dagsenter, Larvik
  - Husebyjordet dagsenter, Lillestrøm
  - Åråsveien dagsenter, Lillestrøm
  - Myraveien Dagsenter, Moss
  - Skogbrynet dagsenter, Moss
  - Dagsenter Nedre Eiker, Nedre Eiker
  - Nes Dagsenter, Nes
  - Bjønnesåsen Dagsenter, Nøtterøy
  - Bjørkås dagsenter, Oppegård
  - Re Dagsenter, Re
  - Sandetun dagsenter, Sande
  - Lunden dagsenter, Sandefjord
  - Sørvald dagsenter, Sørum
  - Eik dagsenter, Tønsberg
  - Nes dagsenter, Tønsberg

REFERENCES:
- [Derived] Olsen C, Pedersen I, Bergland A, Enders-Slegers MJ, Ihlebaek C. Effect of animal-assisted activity on balance and quality of life in home-dwelling persons with dementia. Geriatr Nurs. 2016 Jul-Aug;37(4):284-91. doi: 10.1016/j.gerinurse.2016.04.002. Epub 2016 May 4. PMID 27155968